CLINICAL TRIAL: NCT03363035
Title: Safety and Efficacy of Low Molecular Weight Heparin Versus Rivaroxaban in Chinese Patients Hospitalized With Acute Coronary Syndrome(H-REPLACE): a Prospective, Randomized, Open-label, Active-controlled, Multicenter Trial
Brief Title: Safety and Efficacy of LMWH Versus Rivaroxaban in Chinese Patients Hospitalized With Acute Coronary Syndrome
Acronym: H-REPLACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Shenghua Zhou, Professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-REPLACE-201711
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Myocardial Ischemia; Unstable Angina
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Myocardial Ischemia; Angina, Unstable | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rivaroxaban 2.5 mg (Experimental): One 2.5 mg rivaroxaban tablet twice daily
  Interventions: Drug: Rivaroxaban 2.5 mg
- Rivaroxaban 5 mg (Experimental): One 5 mg rivaroxaban tablet twice daily
  Interventions: Drug: Rivaroxaban 5 mg
- enoxaparin (Active Comparator): Enoxaparin 1mg/kg twice daily SC twice daily
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban 2.5 mg — One 2.5 mg rivaroxaban tablet twice daily until hospital discharge or 12 hours before revascularization therapy for a maximum of 8 days.
  Other Names: Xarelto
  Arms: Rivaroxaban 2.5 mg
Drug: Rivaroxaban 5 mg — One 5 mg rivaroxaban tablet twice daily until hospital discharge or 12 hours before revascularization therapy for a maximum of 8 days.
  Other Names: Xarelto
  Arms: Rivaroxaban 5 mg
Drug: Enoxaparin — Enoxaparin 1mg/kg twice daily SC until hospital discharge or 12 hours before revascularization therapy for a maximum of 8 days.
  Other Names: LWMH
  Arms: enoxaparin

SUMMARY:
H-REPLACE trial is a prospective, randomized, open-label, active-controlled, multicenter study in participants with ACS (STEMI or NSTEMI, unstable angina). All eligible participants receiving background treatment of aspirin plus clopidogrel or ticagrelor will be randomly assigned to either oral rivaroxaban 2.5 mg twice daily or rivaroxaban 5 mg twice daily or subcutaneous (SC) enoxaparin 1mg/kg twice daily until hospital discharge or 12 hours before revascularization therapy for a maximum of 8 days.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is a serious and life threatening condition. Anticoagulation during the acute phase of ACS is effective in reducing ischaemic events. The combination regimen of anticoagulation with dual antiplatelet therapy (DAPT) strategy is more effective than either treatment alone. The most widely used parenteral anticoagulation agent in ACS patients is enoxaparin (1 mg/kg administered subcutaneously twice daily).

Rivaroxaban is a novel oral anticoagulant with potent anti-Xa activity, which might be an attractive alternative drug to enoxaparin. In fact, rivaroxaban was consistently shown to be non-inferior to enoxaparin therapy aimed to reduce the event of recurrent venous thromboembolism. Moreover, the bleeding risk of low dose of rivaroxaban is low and acceptable (1.0-2.5%) during the acute phase of ACS as shown by ATLAS ACS-TIMI 46 Trial, and the bleeding risk of enoxaparin during the acute phase of ACS was 4.3% as shown in a meta-analysis.

We thus hypothesized that the safety and efficacy of rivaroxaban during the acute phase of ACS is non-inferior to enoxaparin and designed this prospective, randomized, open-label, active-controlled, multicenter study in participants with ACS (STEMI or NSTEMI or unstable angina). All eligible participants receiving background treatment of aspirin plus clopidogrel or ticagrelor will be randomly assigned to either receive oral rivaroxaban 2.5 mg twice daily or oral rivaroxaban 5 mg twice daily or enoxaparin 1mg/kg twice daily SC until hospital discharge or 12 hours before revascularization therapy for a maximum of 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Diagnosed with ACS (STEMI, NSTEMI, unstable angina)
* With an indication for short-term combination use of DAPT and enoxaparin.

Exclusion Criteria:

* Already received thrombolytic therapy or revascularization or needing revascularization therapy in 12 hours.
* With platelet glycoprotein IIb/IIIa receptor antagonist therapy.
* With increased bleeding risk, such as but not limited to, active internal bleeding, clinically significant bleeding, bleeding at a non-compressible site, or bleeding diathesis within 30 days of randomization; platelet count less than 90,000/μL at screening; intracranial hemorrhage; major surgery, biopsy of a parenchymal organ, or serious trauma within 30 days before randomization; clinically significant gastrointestinal bleeding within 12 months before randomization; an international normalized ratio known to be>1.5 at the time of screening; abciximab bolus or infusion within the preceding 8 hours, or an eptifibatide or tirofiban bolus or infusion within the past 2 hours preceding randomization; or any other condition known to increase the risk of bleeding.
* Severe concomitant condition or disease, such as cardiogenic shock at the time of randomization, ventricular arrhythmia refractory to treatment at the time of randomization, calculated creatinine clearance b 30 mL/min at screening, known significant liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis), or liver function test abnormalities (confirmed with repeat testing) which would require study drug discontinuation, i.e., aminoleucine transferase (ALT) >5 × the upper limit of the normal range (ULN) or ALT >3 × ULN plus total bilirubin >2 × ULN, prior ischemic stroke or transient ischemia attack, anemia (i.e., hemoglobin < 10 g/ dL＝ at screening, known clinical history of human immunodeficiency virus infection at screening, substance abuse (drug or alcohol) problem within the previous 6 months or any severe condition such as cancer that would limit life expectancy to less than 6 months.
* With an indication for long-term oral anticoagulation therapy such as atrial fibrillation, venous thromboembolism, or prior placement of a mechanical heart valve.
* With other contraindications for use of rivaroxaban and enoxaparin.
* Enrolled in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2055 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Primary Safety Outcome: The percentage of patients with minor, clinically relevant non-major (CRNM) and major bleeding [International Society on Thrombosis and Haemostasis (ISTH) definition of bleeding] | From the time of randomization (Day 1) up to completion of the follow up phase (Month 6)
  The percentage of patients with the first occurrence of bleeding event according to ISTH definition. The statistical analysis was based on the occurrence of the bleeding event from randomization to Month 6.
Primary Efficacy Outcome: The percentage of patients with the composite endpoint of cardiac death, myocardial infarction, re-revascularization or stroke. | From the time of randomization (Day 1) up to completion of the follow up phase (Month 6).
  The percentage of patients with the first occurrence of the composite of death, myocardial infarction, re-revascularization or stroke. The statistical analysis was based on the time from randomization to the first occurrence of the event up to Month 6.

SECONDARY OUTCOMES:
The percentage of patients with the cardiac-related rehospitalization. | From the time of randomization (Day 1) up to completion of the follow up phase (Month 6).
  The percentage of patients with the cardiac-related rehospitalization. The statistical analysis was based on the time from randomization to the first occurrence of the event up to Month 6.
The percentage of patients with the all-cause death. | From the time of randomization (Day 1) up to completion of the follow up phase (Month 6).
  The percentage of patients with the all-cause death. The statistical analysis was based on the time from randomization to the first occurrence of the event up to Month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Shenghua Zhou, Ph.D., Principal Investigator — Second Xiangya Hospital of Central South University
Locations (24):
- China (24):
  - The First People's Hospital of Changde City, Changde, Hunan
  - Changsha Central Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital, The First Affiliated Hospital of Hunan Normal University, Changsha, Hunan
  - The Forth Hospital of Changsha, Changsha, Hunan
  - The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Hospital of Changsha, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Hospital of Changsha, Changsha, Hunan
  - The Second People's Hospital of Hunan Province, Changsha, Hunan
  - The First People's Hospital of Chenzhou, Chenzhou, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - The Second Affiliated Hospital of University of South China, Hengyang, Hunan
  - The First Affiliated Hospital of Hunan University of Medicine, Huaihua, Hunan
  - The First People's Hospital of Huaihua, Huaihua, Hunan
  - The First Affiliated Hospital of Jishou University, Jishou, Hunan
  - The First People's Hospital of Loudi, Loudi, Hunan
  - The Central Hospital of Shaoyang, Shaoyang, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Xiangxiang People's Hospital, Xianxiang, Hunan
  - Yiyang Central Hospital, Yiyang, Hunan
  - Yongzhou First People's Hospital, Yongzhou, Hunan
  - The First People's Hospital of Yueyang, Yueyang, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Q, Ding H, Dai Z, Yang R, Zhou S, Tai S. U-shaped association between plasma cyclic guanosine monophosphate-adenosine monophosphate (cGAMP) levels and myocardial infarction. BMC Cardiovasc Disord. 2025 Feb 19;25(1):116. doi: 10.1186/s12872-025-04543-9. PMID 39972291
- [Derived] Zhou S, Xiao Y, Zhou C, Zheng Z, Jiang W, Shen Q, Zhu C, Pan H, Liu C, Zeng G, Ge L, Zhang Y, Ouyang Z, Fu G, Pan G, Chen F, Huang L, Liu Q; H-REPLACE Investigators. Effect of Rivaroxaban vs Enoxaparin on Major Cardiac Adverse Events and Bleeding Risk in the Acute Phase of Acute Coronary Syndrome: The H-REPLACE Randomized Equivalence and Noninferiority Trial. JAMA Netw Open. 2023 Feb 1;6(2):e2255709. doi: 10.1001/jamanetworkopen.2022.55709. PMID 36763358
- [Derived] Xiao Y, Tang L, Liu Q, Hu X, Fang Z, Zhou S. Rationale and Design of the H-REPLACE Study: Safety and Efficacy of LMWH Versus Rivaroxaban in ChinEse Patients HospitaLized with Acute Coronary SyndromE. Cardiovasc Drugs Ther. 2022 Feb;36(1):69-73. doi: 10.1007/s10557-020-07076-9. Epub 2020 Sep 23. PMID 32965585